CLINICAL TRIAL: NCT02088879
Title: Physical Workload Identify in Chest Compression Position Using Surface Electromyogram
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hanyang University (Other)
Responsible Party: Principal Investigator, Jaehoon Oh, Department of Emergency Medicine, Hanyang University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: EMG CPR-freq1
Record Dates: First submitted 2014-03-13; First posted 2014-03-17 (Estimated); Last update posted 2014-04-02 (Estimated); Status verified 2014-04

CONDITIONS: Cardiopulmonary Resuscitation; Cardiac Arrest
MeSH Terms: conditions — Heart Arrest | interventions — Standing Position

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group1 (Experimental): * first : chest compression with kneeling position
  * second : chst compression with standing position
  Interventions: Behavioral: chest compression with kneeling position; Behavioral: chest compression with standing position
- Group2 (Experimental): * first : chest compression with standing position
  * second : chst compression with kneeling position
  Interventions: Behavioral: chest compression with kneeling position; Behavioral: chest compression with standing position

INTERVENTIONS:
Behavioral: chest compression with kneeling position
Behavioral: chest compression with standing position

SUMMARY:
The chest compression depth decreases over time after starting continuous chest compression due to the rescuers' fatigue.

The investigators hypothesized that the frequency parameters from surface electromyogram from each muscle during chest compression may reflect the muscle fatigue of the rescuers.

Then investigators can identify which of the body are mainly used and get tired by continuous chest compression using surface electromyogram.

ELIGIBILITY:
Inclusion Criteria:

* doctors with American Heart Association Basic Life Support (AHA BLS) provider certification
* healthy, experienced health-care providers

Exclusion Criteria:

* physical pain (ex. low back, wrist)
* heart disease

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2014-03; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
median frequency of electromyogram | two weeks
  median frequency of electromyogram in 16 muscles during chest compression
  The muscles are flexor carpi radialis, extensor carpi radialis, biceps brachii, triceps brachii, deltoideus, erector spinae (cervical area), trapezius, rhomboid, erector spinae (thoracic area), erector spinae (lumbar), obliquus externus abdominis, rectus abdominis, pectoralis, quadriceps femoris, biceps femoris, gastrocnemius. On the dominant side of the rescuers, we will attach sixteen electrodes on these muscles.

CONTACTS AND LOCATIONS:
Overall Officials: Wonhee Kim, M.D., Principal Investigator — Department of emergency medicine, college of medicine, Hanyang university
Locations (1):
- Hanyang University Seoul Hospital, Seoul, South Korea

REFERENCES:
- [Derived] Cho Y, Lee Y, Lim TH, Chee Y, Oh J, Kim W, Jang SH, Kim SM. What muscles need to be trained for high-quality chest compression? Australas Emerg Care. 2020 Dec;23(4):272-280. doi: 10.1016/j.auec.2020.06.002. Epub 2020 Jul 7. PMID 32646835